CLINICAL TRIAL: NCT02935465
Title: Effects of Behavioral Interventions on Mechanisms of Pain Regulation and Hedonic Regulation in Opioid-Treated Chronic Pain Patients
Brief Title: Effects of Behavioral Interventions on Mechanisms of Pain Regulation and Hedonic Regulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Synthesis of the chemical precursor for the neuroimaging radiotracer could not be produced in a stable fashion.
Sponsor: University of Utah (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Eric Garland, Associate Director of Integrative Medicine in Supportive Oncology and Survivorship, Huntsman Cancer Institute; Associate Dean for Research and Associate Professor, College of Social Work, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00093561
Record Dates: First submitted 2016-10-11; First posted 2016-10-17 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Chronic, Non-neuropathic Back Pain
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-Oriented Recovery Enhancement (Experimental): Participants will attend a Mindfulness-Oriented Recovery Enhancement (MORE) group weekly for eight weeks.
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE)
- Support Group (Active Comparator): Participants will attend a support group weekly for eight weeks.
  Interventions: Behavioral: Support Group

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE) — Mindfulness-Oriented Recovery Enhancement (MORE) is a group behavioral intervention that unites mindfulness training, cognitive reappraisal, and positive psychological principles into an integrative intervention strategy targeting mechanisms of pain and opioid misuse.
  Arms: Mindfulness-Oriented Recovery Enhancement
Behavioral: Support Group — A conventional support group will allow participants to express emotions, share experiences, and receive social support under the guidance of a skilled therapist.
  Arms: Support Group

SUMMARY:
The overarching aim of this project is to conduct a randomized controlled study to determine whether Mindfulness-Oriented Recovery Enhancement (MORE) vs. a Support Group (SG) can improve pain regulation and hedonic functions (i.e., natural reward responsiveness) thought to be governed by the endogenous opioid system among opioid-treated, chronic, non-neuropathic back pain patients (CNBP) and thereby improve clinical pain, affect, and opioid use.

ELIGIBILITY:
Inclusion Criteria:

1. age 21-60 years of age
2. English fluency
3. 20/20 vision with corrective lenses
4. current chronic, non-neuropathic back pain diagnosis determined by physician assessment
5. reporting pain ≥3 on 0-10 scale with opioid medication
6. current use of prescription opioids for ≥3 consecutive months
7. ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

1. Mindfulness experience (e.g., MBSR or shamatha/vipassana meditation)
2. psychosis
3. untreated, active suicidality in the past month
4. and severe non-opioid substance use disorder in the past year as assessed with the MINI
5. clinically unstable illness judged to interfere with treatment, and presence of facial/jaw pain
6. pregnancy
7. inability or unwillingness of individual to give written informed consent
8. physical characteristics that preclude neuroimaging or study procedures (e.g., metal implants, etc.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Changes in endogenous opioid system function in response to pain challenge | Change from week 0 to 8 weeks
  PET opioid receptor binding potential from baseline through pain challenge
Changes in fMRI activity level during natural reward processing | Change from week 0 to 8 weeks
  Blood oxygen dependent signal (BOLD) response during viewing and regulating response to natural reward cues measured during a fMRI scan.

SECONDARY OUTCOMES:
Pain sensitivity as a measure of volume of hypertonic saline | Change from week 0 to 8 weeks
  Volume of hypertonic saline to maintain pain at 40 out of 100 on a VAS
Self-report affect ratings | Change from week 0 to 8 weeks
Significant correlation between PET and fMRI measures with improvements in clinical pain, affect, and opioid use | Change from week 0 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Garland, PhD, Principal Investigator — The University of Utah
Locations (1):
- College of Social Work, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided